CLINICAL TRIAL: NCT05013489
Title: Physicians Burnout: Cause, Consequence and Mindfulness and Intercare Based Intervention for Physicians Burnout Reduction
Brief Title: Mindfulness and Intercare Based Intervention for Physicians Burnout Reduction
Acronym: MIIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Diego Portales (Other)
Responsible Party: Principal Investigator, Francisco Javier Villalon Lopez, Principal Investigator, University Diego Portales
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-2020
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Burnout; Mental Health Wellness 1
MeSH Terms: conditions — Burnout, Psychological | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness, compassion and intercare based Intervention (Experimental): An Eight week mindfulness and intercare group online program.
  Interventions: Behavioral: Mindfulness and intercare based intervention
- Waiting list (No Intervention): Psychological support if needed. No other intervention.

INTERVENTIONS:
Behavioral: Mindfulness and intercare based intervention — Eight week online program based on mindfulness, compassion and intercare intervention. A two hour synchronic online session every week plus daily homework based on meditation and journaling exercises.
  The topics covered in the program are mindfulness meditation, cognitive behavioral therapy exercises, gratitude and acceptance, compassion and self compassion exercises, conservation of resources theory and intercare.
  Arms: Mindfulness, compassion and intercare based Intervention

SUMMARY:
During the coronavirus disease 2019 (COVID19) pandemic, many physicians have presented burnout. A range of associated factors need to be considered for effective prevention and intervention. Objective 1: To assess the association of burnout in medical doctors with individual factors, self-reported medical errors, medical leave, and demands of the work environment demand. Objective 2: to assess the effectiveness of a online mindfulness, compassion and intercare based intervention to reduce burnout.

ELIGIBILITY:
Inclusion Criteria:

* Physicians enrolled in the database of the medical college of Chile

Exclusion Criteria:

* Recent Grief
* Severe acute depression disorder
* Active suicidal ideation
* Active Psychosis
* Active addiction
* Post Traumatic Stres Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, female, Other
Enrollment: 795 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Maslach Burnout Inventory - Human Services | Baseline
  Burnout was evaluated with Maslach Burnout Inventory for Human Services. Continuous variable for burnout total score, emotional exhaustion, depersonalization and accomplishment. Dichotomous variable was used for burnout syndrome using two common cut-off point criteria and a new proposal.
Maslach Burnout Inventory - Human Services | 3 months
  Burnout was evaluated with Maslach Burnout Inventory for Human Services. Continuous variable for burnout total score, emotional exhaustion, depersonalization and accomplishment. Dichotomous variable was used for burnout syndrome using two common cut-off point criteria and a new proposal.
Maslach Burnout Inventory - Human Services | 6 months
  Burnout was evaluated with Maslach Burnout Inventory for Human Services. Continuous variable for burnout total score, emotional exhaustion, depersonalization and accomplishment. Dichotomous variable was used for burnout syndrome using two common cut-off point criteria and a new proposal.

SECONDARY OUTCOMES:
Demands of the work environment - Psychosocial Factors Questionnaire 75. (PFQ-75-SF) | Baseline
  Demands of the work environment were evaluated with an adaptation of the Psychosocial Factors Questionnaire 75.
Demands of the work environment - Psychosocial Factors Questionnaire 75. (PFQ-75-SF) | 3 months
  Demands of the work environment were evaluated with an adaptation of the Psychosocial Factors Questionnaire 75.
Demands of the work environment - Psychosocial Factors Questionnaire 75. (PFQ-75-SF) | 6 months
  Demands of the work environment were evaluated with an adaptation of the Psychosocial Factors Questionnaire 75.
Medical error perception - Medical Error Checklist General (MECG) | Baseline
  Medical error perception was evaluated with an adaptation of the Medical Error Checklist.
Medical error perception - Medical Error Checklist General (MECG) | 3 months
  Medical error perception was evaluated with an adaptation of the Medical Error Checklist.
Medical error perception - Medical Error Checklist General (MECG) | 6 months
  Medical error perception was evaluated with an adaptation of the Medical Error Checklist.
Medical Leave | Baseline
  Days of medical leave if needed
Medical Leave | 3 months
  Days of medical leave if needed
Medical Leave | 6 months
  Days of medical leave if needed
Personality - The Big Five Inventory-2 Short Form (BFI-2-S) | Baseline
  As individual factors were measured Personality with a short version of the Big Five Questionnaire The Big Five Inventory-2 Short Form (BFI-2-S)
Mental Health - Mental Health Continuum Scale- Short Form | Baseline
  Mental Health - Mental Health Continuum Scale- Short Form (MHC-14): Mental health can be defined as a state in which an individual realizes his or her own abilities, can cope with the stresses of life, can work productively and can make a contribution,and is described by Corey L. Keyes in 3 main dimensions; emotional well being, psychological well being and social well being.
  It is a Likert from 0 to 5 with a total of 14 ítems and 3 main subdimensions: emotional well being (BE, 3 ítems), psychological well being (BP, 5 ítems) y social well being.(PS, 6 ítems). It as a total score of 70 and a minium of 0. The higher the better mental health.
Mental Health - Mental Health Continuum Scale- Short Form | 3 months
  Mental Health - Mental Health Continuum Scale- Short Form (MHC-14): Mental health can be defined as a state in which an individual realizes his or her own abilities, can cope with the stresses of life, can work productively and can make a contribution,and is described by Corey L. Keyes in 3 main dimensions; emotional well being, psychological well being and social well being.
  It is a Likert from 0 to 5 with a total of 14 ítems and 3 main subdimensions: emotional well being (BE, 3 ítems), psychological well being (BP, 5 ítems) y social well being.(PS, 6 ítems). It as a total score of 70 and a minium of 0. The higher the better mental health.
Mental Health - Mental Health Continuum Scale- Short Form | 6 months
  Mental Health - Mental Health Continuum Scale- Short Form (MHC-14): Mental health can be defined as a state in which an individual realizes his or her own abilities, can cope with the stresses of life, can work productively and can make a contribution,and is described by Corey L. Keyes in 3 main dimensions; emotional well being, psychological well being and social well being.
  It is a Likert from 0 to 5 with a total of 14 ítems and 3 main subdimensions: emotional well being (BE, 3 ítems), psychological well being (BP, 5 ítems) y social well being.(PS, 6 ítems). It as a total score of 70 and a minium of 0. The higher the better mental health.
Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) | Baseline
  Mindfulness is defined as the ability to pay attention to our own experiences without judging them. The Five Facet Mindfulness Questionnaire Short Form was used, which consists of 24 questions that look for the 5 facets of mindfulness: observe, describe, act aware, non-judge and no-react.
Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) | 3 months
  Mindfulness is defined as the ability to pay attention to our own experiences without judging them. The Five Facet Mindfulness Questionnaire Short Form was used, which consists of 24 questions that look for the 5 facets of mindfulness: observe, describe, act aware, non-judge and no-react.
Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) | 6 months
  Mindfulness is defined as the ability to pay attention to our own experiences without judging them. The Five Facet Mindfulness Questionnaire Short Form was used, which consists of 24 questions that look for the 5 facets of mindfulness: observe, describe, act aware, non-judge and no-react.
Self compassion scale Short form (SCS-SF) | Baseline
  Self compassion is understood as maintenance of full attention and opening without disconnecting from self's suffering with the desire to alleviate it in a non judgemental way, comprehending the own experience as a part of the human experience. The "Self Compassion Scale Short Form - 12 a scale of 6 sub domains was used.
Self compassion scale Short form (SCS-SF) | 3 months
  Self compassion is understood as maintenance of full attention and opening without disconnecting from self's suffering with the desire to alleviate it in a non judgemental way, comprehending the own experience as a part of the human experience. The "Self Compassion Scale Short Form - 12 a scale of 6 sub domains was used.
Self compassion scale Short form (SCS-SF) | 6 months
  Self compassion is understood as maintenance of full attention and opening without disconnecting from self's suffering with the desire to alleviate it in a non judgemental way, comprehending the own experience as a part of the human experience. The "Self Compassion Scale Short Form - 12 a scale of 6 sub domains was used.

CONTACTS AND LOCATIONS:
Locations (1):
- University Diego Portales, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Villalon Lopez F, Mundt AP, Hirmas A, Rivera RM, Guiloff R. Impact of burnout on turnover, medical errors, medical leave and a cross-sectional study of contributing factors among Chilean physicians. BMJ Open. 2025 May 15;15(5):e099773. doi: 10.1136/bmjopen-2025-099773. PMID 40379332